CLINICAL TRIAL: NCT00225121
Title: A PHASE 1, OPEN-LABEL, DOSE-ESCALATION STUDY TO EVALUATE SAFETY, PHARMACOKINETICS AND PHARMACODYNAMICS OF 2 DOSING SCHEDULES OF PF-00299804 IN PATIENTS WITH ADVANCED MALIGNANT SOLID TUMORS
Brief Title: Study To Evaluate The Safety, Pharmacokinetics, And Pharmacodynamics Of PF-00299804 In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A7471001; 2005-001140-23 (EudraCT Number); NCT00276653 (obsolete NCT alias); NCT00278291 (obsolete NCT alias)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): open label single arm trial
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — investigational drug by oral route (escalating doses depending on safety) administered until progression

SUMMARY:
The primary purpose of this study is to study the side effects of PF-00299804 and determine the highest dose that can be safely administered in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Malignant solid tumor for which there is no currently approved treatment
* Adequate bone marrow, liver, cardiac, and kidney function

Exclusion Criteria:

* Cardiac disease
* Anticancer therapy within 4-6 weeks (depending on therapy)
* Pregnant or breast-feeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-10-11 (Actual); Primary Completion 2007-04-03 (Actual); Study Completion 2010-09-23 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months

SECONDARY OUTCOMES:
Pharmacokinetics | 6 months
Pharmacodynamics | 6 months
Efficacy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (8):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Oncology Center, Los Angeles, California
  - UCLA Hematology Oncology - Santa Monica, Santa Monica, California
  - UCLA Santa Monica Hematology/Oncology, Santa Monica, California
  - University of Colorado Hospital, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
- Vereniging het Nederlandse Kanker Instituut, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Janne PA, Boss DS, Camidge DR, Britten CD, Engelman JA, Garon EB, Guo F, Wong S, Liang J, Letrent S, Millham R, Taylor I, Eckhardt SG, Schellens JH. Phase I dose-escalation study of the pan-HER inhibitor, PF299804, in patients with advanced malignant solid tumors. Clin Cancer Res. 2011 Mar 1;17(5):1131-9. doi: 10.1158/1078-0432.CCR-10-1220. Epub 2011 Jan 10. PMID 21220471
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471001&StudyName=Study%20To%20Evaluate%20The%20Safety%2C%20Pharmacokinetics%2C%20And%20Pharmacodynamics%20Of%20PF-00299804%20In%20Patients%20With%20Advanced%20Solid%20Tumors